CLINICAL TRIAL: NCT02614378
Title: Abortive Effect of an Ear Insufflator on Migraine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carrick Institute for Graduate Studies (Other)
Responsible Party: Principal Investigator, Frederick Carrick, PhD, FACCN, Principal Investigator, Carrick Institute for Graduate Studies
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CI-IRB-20151104001
Record Dates: First submitted 2015-11-21; First posted 2015-11-25 (Estimated); Last update posted 2016-12-14 (Estimated); Status verified 2016-12

CONDITIONS: Migraine
Keywords: abortive effect
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Subject receiving treatment (Active Comparator): participant receiving air insufflation
  Interventions: Procedure: air insufflation
- Subject receiving placebo (Placebo Comparator): participant not receiving air insufflation
  Interventions: Procedure: placebo

INTERVENTIONS:
Procedure: air insufflation — modulated air insufflation of the ear canal
  Arms: Subject receiving treatment
Procedure: placebo — no air will be introduced in the ear canal
  Arms: Subject receiving placebo

SUMMARY:
Evaluate the effectiveness of air insufflation in aborting (stopping) an acute episode of migraine and compare it with a placebo effect of using the same procedure but without active insufflation. The insufflation will be used when the subject is experiencing an acute episode of migraine to determine its ability to reduce, if not to completely eliminate the migraine symptoms. Subjects receiving the placebo treatment will be offered the active treatment during the subsequent episode of migraine.

DETAILED DESCRIPTION:
Each patient will be asked (using a questionnaire) to describe the nature of their presenting symptoms including distribution pattern, symmetry, laterality, severity and associated symptoms. Severity of migraine/headache will be recorded. The patient's description of their symptoms will be used to guide the treatment process in terms of treatment time and side (i.e. left or right ear). A tubular soft silicone ear-plug will be inserted into the patient's ear on the side of greatest reported severity. In the absence of clear laterality with respect to severity, the side associated with the greatest surface area of involvement will be selected (e.g., the patient has a bilateral headache but on the left, it is perceived as retro-orbital whereas on the right it is retro-orbital and temporal, therefore the right side will be selected), In the absence of lateralizing features, the initial treatment side will be randomly selected. Then the air insufflation will start. The patient will be encouraged to relax during the process and the extent of the insufflation will be maintained a level that is comfortable for the patient. The patient will be asked to report any sense of aggravation of their symptoms, which would prompt the examiner to suspend the treatment. The patient will not know if the treatment received is the active or the placebo one.

Following insufflation, the ear plug will be removed and the patient will be asked to rate the severity of their symptoms and describe any changes in characteristics. A significant reduction in pain level will be considered an indication that the treatment is appropriate for that patient and the treatment will then continue on the ipsilateral side. If the patients will describe resolution of their symptoms in a hemi-distribution of the head ("the symptoms are gone from this side of my head but they're still left on the other side"), the treatment process will be repeated on the contralateral side until resolution (or maximal reduction in symptoms) will be achieved. Treatment session in this study will last 20 minutes.

There will be a followup at 2h and 24h post treatment to monitor the status of the patient and they will all be invited back for a second treatmentduring the subsequent episode of migraine.

Vitals (blood pressure, heart rate, pulse oxygenation and temperature) will also be monitored to see if there are any changes before and immediately after treatment.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects suffering from acute migraine episodes
* Possibly located in the Phoenix, AZ area

Exclusion Criteria:

* Pregnant/nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Changes in Symptoms severity scale | pre-treatment, immediately post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and immediately post treatment

SECONDARY OUTCOMES:
Changes in Symptoms severity scale at 2h | pre-treatment, 2h post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and 2h post treatment
Changes in Symptoms severity scale at 24h | pre-treatment, 24h post-treatment
  Subjects will grade the severity of their symptoms on a scale from 0 to 10. Changes in the symptoms severity scale will be assessed between pre and 24h post treatment
Changes in blood pressure | pre-treatment, immediately post-treatment
  Blood pressure will be measured. Changes in blood pressure will be assessed between pre and immediately post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Frederick R Carrick, PhD, Principal Investigator — Carrick Institute for Graduate Studies
Locations (2):
- United States (2):
  - Buckler Chiropractic, Phoenix, Arizona
  - Doctor's office, Scottsdale, Arizona

IPD SHARING:
Plan to Share IPD: No